CLINICAL TRIAL: NCT00065728
Title: An Open Label Evaluation of Long Term Efficacy and Safety of Posterior Juxtascleral Injections of Anecortave Acetate 15 mg in Patients With Subfoveal Exudative Age-Related Macular Degeneration (AMD)
Brief Title: Open-Label Posterior Juxtascleral Injections of Anecortave Acetate 15mg Dose for Long Term Use in Patients With AMD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-03-15
Record Dates: First submitted 2003-07-31; First posted 2003-08-01 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2009-05

CONDITIONS: Macular Degeneration
Keywords: AMD; age-related macular degeneration; Anecortave; Acetate; Wet form of age-related macular degeneration; CNV; Anecortave Acetate
MeSH Terms: conditions — Macular Degeneration | interventions — anecortave acetate; AL 3789

ARMS (1):
- Anecortave Acetate, 15 mg (Experimental): One 0.5 mL injection of 30 mg/mL Anecortave Acetate sterile suspension into the posterior juxtascleral depot at 6 month intervals for 18 months
  Interventions: Drug: Anecortave Acetate (AL-3789) Sterile Suspension, 30 mg/mL

INTERVENTIONS:
Drug: Anecortave Acetate (AL-3789) Sterile Suspension, 30 mg/mL — One 0.5 mL injection of 30 mg/mL Anecortave Acetate sterile suspension into the posterior juxtascleral depot at 6 month intervals for 18 months

SUMMARY:
The purpose of this study is to investigate the long-term efficacy and safety of posterior juxtascleral injections of open label Anecortave Acetate 15mg administered every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subfoveal exudative age-related macular degeneration (AMD) who were previously enrolled in long-term studies with anecortave acetate.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2003-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Percent of patients who maintained stable vision | Month 24
  Stable vision is defined as < 15-letter loss of best-corrected visual acuity scores)
Mean change in best-corrected visual acuity at Month 24 from baseline | Baseline, Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Terry Wiernas, PhD, Study Director — Alcon Research
Locations (1):
- Belgium,France,Germany,Hungary,Italy,Netherlands,Poland,Spain,Sweden,UK, Central Contact Fort Worth, Texas, United States